CLINICAL TRIAL: NCT04276766
Title: Exploring the Effect of Inorganic Nitrates on the Human Microvascular Physiology - a Pilot Study.
Acronym: ENIH-MPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: University of Sheffield (Other); University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: HWB-S&E-23
Record Dates: First submitted 2020-02-13; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Aging
Keywords: nitrates; beetroot; nutrition; microcirculation; nitrites

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beetroot (Experimental): Following baseline microcirculatory and blood pressure measurements, as well as the collection of urine and saliva samples, participants on the "beetroot" group were asked to consume 140ml beetroot juice (James White Drinks Company, Suffolk, UK). The 140 ml of beetroot juice equate to approximately 8.4 mmol of NO3- .
  Interventions: Other: Crossover intervention
- Placebo (Placebo Comparator): Following baseline microcirculatory and blood pressure measurements, as well as the collection of urine and saliva samples, participants on the "placebo" group were asked to consume 140 ml nitrate-depleted beetroot juice (James White Drinks Company, Suffolk, UK).
  Interventions: Other: Crossover intervention

INTERVENTIONS:
Other: Crossover intervention — Drink consumption was followed by regular BP measurements and collection of saliva samples every 30 minutes for four hours. Microcirculatory measurements were then repeated and saliva and urine samples were collected again.
  After the last measurement subjects were provided with a standardized meal with a very low nitrate intake to eat within 30minutes. Participant then left the research centre and they were asked to collect a saliva sample after two hours from the completion of the meal. This was immediately followed a dose of labelled nitrate (4mg in 100ml of distilled water) to drink within one minute. Subjects were then asked to collect six additional saliva samples until the next morning (four before going to bed and two in the morning), accompanied by measurements of resting BP.
  Cross-over assessments were then repeated in the same order at Visit 3, followed a wash-out period of at least one week before entering the second arm of the study.

SUMMARY:
We conducted a randomised, placebo-controlled, double blind, cross-over, trial to examine the short-term effect of concentrated beetroot juice on vascular outcomes in a young (18-35 years) and older group (55-75 years). The study included a run-in period of one day preceding the test day. A wash-out period of at least 7 days was implemented to ensure to avoid a carry-over effect of the interventions.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the largest cause of global mortality accounting for over twenty-nine percent of all deaths with coronary heart disease and stroke projected to become the global leading causes of mortality by 2020. Increased mortality represents only one side of the problem since the clinical care of CVD is costly and prolonged and potentially diverts family and societal resources towards life-saving intensive medical treatments. Therefore, it is crucial to develop preventative and therapeutic strategies that will reduce the financial and social burden of CVD.

Ageing is a major risk factor for chronic diseases such as cancer, diabetes neurodegeneration and CVD. For example, the prevalence and incidence of Chronic Venous Insufficiency (CVI) is closely linked to an age-related dysfunction of micro-circulation control. Similarly, ageing is associated with increased risk of atherosclerosis and formation of macroscopic lesions in large arteries leading to obstruction of blood flow and onset of ischaemic events . The rapid changes in worldwide trends of age-demographics are therefore closely correlated with the rising burden of CVD.

Hypertension is an important risk factor for CVD. Raised blood pressure (BP) is primarily caused by increased vascular resistance, mainly due to arterial wall thickening, autonomic dysregulation and endothelial dysfunction . Endothelium-derived nitric oxide (NO) is a potent vasodilator that plays a pivotal role in the moment-to-moment control of vascular tone . Therefore, it is no surprise that a key aspect of endothelial dysfunction is a reduced NO production via the L-arginine-dependent enzymatic pathway. NO also decreases platelet aggregation, improves mitochondrial function, and diminishes cellular vascular adhesion . Hence a reduction in NO bioavailability is causally related to an increase in BP and atherosclerotic risk.

Until recently it was believed that dietary nitrate (NO3-) and nitrite (NO2-) offered limited physiological benefits, despite them being produced endogenously as part of the NO metabolic pathway . The discovery of the entero-salivary circulation and non-enzymatic reduction of NO3- into NO2- and NO provides an important alternative source of NO, particularly in environment with reduced pH and oxygen tension . The major sources of dietary NO3- are green leafy vegetables such as rocket or spinach or tuberous product such as beetroot. The typical nitrate intake of a western diet provides between 50-100mg/NO3-/day whereas diets rich in fruit- and vegetables such as the Mediterranean or Japanese diets could provide up to 1000mg/NO3-/day. Increasing evidence seems to support the association between the high NO3- content of these dietary patterns with protective cardiovascular effects.

The cardiovascular benefits of NO3- are thought to be derived by an improvement of endothelial function achieved by improved NO bioavailability. Other mechanisms may include a direct effect of NO2- on calcium-channels in vascular smooth muscle cells (SMVCs) in resistance vessels . The conversion of NO3- into NO2- by the oral micro-environment is a key mechanism of the entero-salivary NO3- circulation and non-enzymatic synthesis of NO. The oral microbiota is critically involved in the first reducing step (NO3- into NO2-) and an alteration of the reducing capacity of the oral microbiota (i.e., spitting, antiseptic mouthwash) interrupts the beneficial effects of inorganic NO3- on vascular function. Siervo et al has recently demonstrated a reduced efficacy of concentrated beetroot juice supplementation in older overweight and obese subjects. Ageing appears to be linked to changes in the oral micro-environment as well as a reduced responsiveness of the endothelium and SMVCs to NO.

However, there is limited knowledge on the influence of the ageing process on factors that affect NO3- conversion starting from the NO3- -reducing potential in the oral environment. Therefore, a better understanding of the age-related mechanisms linked to endothelial dysfunction could lead to the development of effective and targeted dietary strategies for the early prevention of hypertension, arterial stiffness and CVD across the life-course.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking,
* healthy (defined by the absence of overt chronic diseases that could affect their micro- and macro- vascular function - e.g. chronic venous insufficiency, systemic sclerosis, hypercholesterolemia, diabetes, cardiovascular disease - as determined by a medical history questionnaire),
* male or female adults aged between 18 and 35 years (Group A) and 55 and 75 years (Group B).
* normotensive (systolic blood pressure (SBP) between 115 and 140 mmHg and diastolic blood pressure (DBP) between 75 and 90 mmHg) with body mass index (BMI) 18-30 kg/m2.

Exclusion Criteria:

* taking medications interfering with the study outcomes,
* have lost more than 3kg in the month before the study,
* wearing complete dentures and diagnosis of inflammatory oral diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Change of micro-circulatory function from baseline | 3 hours
  Non-invasive laser Doppler flowmetry (LDF) measurements (Periflux 5000 System, Perimed, Sweden) will be used as an index of cutaneous (microcirculatory) function and red blood cell flux. To obtain a measure of microcirculatory, NO-dependent, endothelial-function (26) measurements will be taken once at Visit 1 and twice (prior to and 3 hrs. after beverage ingestion) on Visits 2 and 3, using thermal hyperaemia. For this, four 7-point integrating probes (Model 413, Perimed) housed within local heating units (Model 455, Perimed) will be placed on the ventral aspect of the left forearm. The heating units will be initially set at 33 °C. After a 10-min baseline recording, the temperature of the heating unit will then be increased to 42 °C at a rate of 1 °C every 10 seconds to obtain maximum skin blood flow; this (i.e., a stable plateau in skin blood flow) is usually observed after approx. 25 minutes of localised heating.

SECONDARY OUTCOMES:
Blood pressure measurements | Up to 24 hours
  Resting BP sure will be recorded intermittently throughout the test using an automated system (Dinamap Dash 2500, GE Healthcare. Duplicate measurements of BP wil be performed covertly and only showed to the participant at the end of the study visit. Before each measurement participants will be invited to rest in a sitting position for at least 15 minutes.
Oral nitrate reductase capacity | Up to 24 hours
  Nitrate reductase activity will be investigated by evaluating the differences in salivary nitrite concentrations according to a validated method. Briefly, ten millilitres of a solution of potassium nitrate in distilled water will be held in the mouth for 5 min and then collected. Background levels of nitrate reduction were estimated by subtracting values obtained from holding distilled water alone in the mouth. NO3- and NO2- concentrations will be measured by chemiluminescence.
Whole-body NO production | Up to 24 hours
  A non-invasive stable isotopic method will be used to assess whole-body NO production (ONT Method). Subjects will receive an oral dose of labelled sodium nitrate in 100ml of distilled water (4mg Na15NO3) and the isotopic decay of the tracer in saliva samples will be used to derive estimates of NO production. Nitrate concentrations will be measured by chemiluminescence. Nitrate enrichments will be measured using Gas Chromatography Mass Spectrometry (GCMS).
Urine / saliva sampling | Up to 24 hours
  Mid-stream urine samples will be collected into sterile containers and an aliquot and will stored at -80 ⁰C until analysis at a later date. Saliva will be collected into sterile eppendorfs and stored at -80 ⁰C until analysis at a later date. Both salivary and urinary samples will be used for NO3- and NO2- measurements. Saliva samples will also be used to assess isotopic enrichment of labelled NO3- as previously described. Sodium hydroxide will be added to urine and saliva samples to avoid nitrate degradation.

IPD SHARING:
Plan to Share IPD: No
Due to ethical approval restrictions there were no plans for IPD available to other researchers.